CLINICAL TRIAL: NCT01181128
Title: A-LONG: An Open-Label, Multicenter Evaluation of the Safety, Pharmacokinetics, and Efficacy of Recombinant Factor VIII Fc Fusion Protein (rFVIIIFc) in the Prevention and Treatment of Bleeding in Previously Treated Subjects With Severe Hemophilia A
Brief Title: Study to Evaluate the Safety, Pharmacokinetics and Efficacy of Recombinant Factor VIII Fc Fusion Protein (rFVIIIFc) in Previously Treated Subjects With Severe Hemophilia A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioverativ Therapeutics Inc. (Industry)
Collaborators: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 997HA301
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2021-01-08 (Actual); Status verified 2017-07

CONDITIONS: Severe Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; F8 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Individualized (Tailored) Prophylaxis (Experimental): On rFVIIIFc Day 0, all participants underwent pharmacokinetic (PK) analysis with 50 IU/kg rFVIIIFc to estimate their PK parameters and guide the appropriate dose or interval of dosing. A subset of participants (Sequential PK subgroup) also had PK analyses performed with a single dose of 50 IU/kg Advate (Advate Day 0) within 8 weeks prior to rFVIIIFc Day 0. A >= 96 hour washout was performed before the PK dose of Advate or rFVIIIFc was administered. Repeat PK profiling with a single dose of 50 IU/kg rFVIIIFc was conducted at Week 14 or after 12 to 24 weeks of prophylaxis with rFVIIIFc.
  After PK assessments, all participants started twice weekly treatment with 25 IU/kg of rFVIIIFc via intravenous (IV) injection on Day 1 and 50 IU/kg on Day 4, followed by individualized dose and interval modification within the range of 25 to 65 IU/kg every 3 to 5 days, as determined by rFVIIIFc PK analysis, to maintain a trough level of 1% to 3% (or higher, as clinically indicated) FVIII activity.
  Interventions: Drug: Factor VIII (rFVIIIFc); Drug: Advate®
- Weekly Prophylaxis (Experimental): 65 IU/kg of rFVIIIFc via IV injection every 7 days
  Interventions: Drug: Factor VIII (rFVIIIFc)
- Episodic (On-Demand) Dosing (Experimental): 10 to 50 IU/kg rFVIIIFc via IV injection, as required to treat a bleeding episode
  Interventions: Drug: Factor VIII (rFVIIIFc)

INTERVENTIONS:
Drug: Factor VIII (rFVIIIFc)
  Other Names: Recombinant Factor VIII Fc Fusion Protein
Drug: Advate®
  Other Names: octocog alfa; Antihemophilic Factor [Recombinant] Plasma/Albumin Free Method
  Arms: Individualized (Tailored) Prophylaxis

SUMMARY:
The primary objectives of this study are: to evaluate the safety and tolerability of rFVIIIFc administered as a prophylaxis (Arm 1), weekly (Arm 2), on-demand (Arm 3), and surgical treatment regimen; to evaluate the efficacy of the rFVIIIFc tailored prophylaxis regimen (Arm 1); to evaluate the efficacy of rFVIIIFc administered as an on-demand (Arm 3) and surgical treatment regimen. The secondary objectives of this study are: to characterize the PK profile of rFVIIIFc and compare the PK of rFVIIIFc with the currently marketed product, Advate®; to characterize the range of dose and schedules required to adequately prevent bleeding in a prophylaxis regimen, maintain hemostasis in a surgical setting, or to treat bleeding episodes in an on-demand, weekly treatment, or prophylaxis setting.

DETAILED DESCRIPTION:
Participants are assigned to one of three treatment regimens: 1) a tailored prophylaxis regimen, 2) a weekly dosing regimen, or 3) an on-demand regimen. Treatment continued for 28 (±2) to 52 (±2) weeks. PK assessments for all participants are conducted on varying schedules, according to participants' group assignments. Additionally, two subgroups are defined. One subgroup of participants undergo PK profiling with a single dose of the comparator Advate®. A second subgroup consists of participants from any of the treatment arms that required surgery during the study. Depending upon country location, participants might have the option of continuing treatment within study 8HA01EXT (NCT01454739).

ELIGIBILITY:
Inclusion Criteria:

* Male, ≥12 years of age with weight at least 40 kg
* Diagnosed with severe hemophilia A, defined as <1 IU/dL (<1%) endogenous Factor VIII)
* History of at least 150 documented prior exposure days to any Factor VIII product
* Platelet count ≥100,000 cells/μL

Exclusion Criteria:

* History of Factor VIII inhibitors
* Kidney and liver dysfunction
* Diagnosed with other coagulation disorder(s) in addition to hemophilia A
* Prior history of hypersensitivity or anaphylaxis associated with any FVIII or IV immunoglobulin administration

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2010-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Bioverativ Therapeutics Inc.
Locations (61):
- United States (20):
  - Research Site, Little Rock, Arkansas
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Indianapolis, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Louisville, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Boston, Massachusetts
  - Research Site, East Lansing, Michigan
  - Research Site, Las Vegas, Nevada
  - Research Site, New York, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Houston, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Seattle, Washington
- Australia (3):
  - Research Site, Camperdown, New South Wales
  - Research Site, Adelaide, South Australia
  - Research Site, Perth, Western Australia
- Research Site, Vienna, Austria
- Research Site, Brussels, Belgium
- Research Site, Campinas, Brazil
- Canada (3):
  - Research Site, Calgary
  - Research Site, Toronto
  - Research Site, Vancouver
- Research Site, Lyon, France
- Germany (2):
  - Research Site, Bonn, Northwest
  - Research Site, Berlin, State of Berlin
- Research Site, Hong Kong, Hong Kong
- India (5):
  - Research Site, Bangalore, Karna
  - Research Site, Pune, Mahara
  - Research Site, New Delhi, National Capital Territory of Delhi
  - Research Site, Ludhiana, Punjab
  - Research Site, Vellore, Tamil Nadu
- Research Site, Ramat Gan, Israel
- Italy (3):
  - Research Site, Florence, FI
  - Research Site, Milan, MI
  - Research Site, Vicenza, VI
- Japan (6):
  - Research Site, Kashihara-shi
  - Research Site, Kawasaki-shi
  - Research Site, Kitakyushu-shi
  - Research Site, Nagoya
  - Research Site, Shinjuku-ku
  - Research Site, Suginami-ku
- New Zealand (3):
  - Research Site, Auckland
  - Research Site, Christchurch
  - Research Site, Palmerston North
- South Africa (2):
  - Research Site, Johannesburg Parktown, Gauteng
  - Research Site, Cape Town, W Cape
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Madrid
- Research Site, Gothenburg, Sweden
- Research Site, Zurich, Switzerland
- United Kingdom (4):
  - Research Site, Basingstoke
  - Research Site, Cambridge
  - Research Site, Glasgow
  - Research Site, London

REFERENCES:
- [Result] Mahlangu J, Powell JS, Ragni MV, Chowdary P, Josephson NC, Pabinger I, Hanabusa H, Gupta N, Kulkarni R, Fogarty P, Perry D, Shapiro A, Pasi KJ, Apte S, Nestorov I, Jiang H, Li S, Neelakantan S, Cristiano LM, Goyal J, Sommer JM, Dumont JA, Dodd N, Nugent K, Vigliani G, Luk A, Brennan A, Pierce GF; A-LONG Investigators. Phase 3 study of recombinant factor VIII Fc fusion protein in severe hemophilia A. Blood. 2014 Jan 16;123(3):317-25. doi: 10.1182/blood-2013-10-529974. Epub 2013 Nov 13. PMID 24227821
- [Result] Shapiro AD, Ragni MV, Kulkarni R, Oldenberg J, Srivastava A, Quon DV, Pasi KJ, Hanabusa H, Pabinger I, Mahlangu J, Fogarty P, Lillicrap D, Kulke S, Potts J, Neelakantan S, Nestorov I, Li S, Dumont JA, Jiang H, Brennan A, Pierce GF. Recombinant factor VIII Fc fusion protein: extended-interval dosing maintains low bleeding rates and correlates with von Willebrand factor levels. J Thromb Haemost. 2014 Nov;12(11):1788-800. doi: 10.1111/jth.12723. Epub 2014 Oct 10. PMID 25196897
- [Derived] Raheja P, Kragh N, Bystricka L, Eriksson D, Aroui K, Mezghani M, Barbier S, Linari S. Long-term efmoroctocog alfa prophylaxis improves perceived pain, mental, and physical health in patients with hemophilia A: post hoc analysis of phase III trials using patient-reported outcomes. Ther Adv Hematol. 2024 Jul 30;15:20406207241257917. doi: 10.1177/20406207241257917. eCollection 2024. PMID 39091324
- [Derived] Katragadda S, Neelakantan S, Diao L, Wong N. Population Pharmacokinetic Analysis of Recombinant Factor VIII Fc Fusion Protein in Subjects With Severe Hemophilia A: Expanded to Include Pediatric Subjects. J Clin Pharmacol. 2021 Jul;61(7):889-900. doi: 10.1002/jcph.1854. Epub 2021 Apr 14. PMID 33719084

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Individualized (Tailored) Prophylaxis: On rFVIIIFc Day 0, all participants underwent pharmacokinetic (PK) analysis with 50 IU/kg rFVIIIFc to estimate their PK parameters and guide the appropriate dose or interval of dosing. A subset of participants (Sequential PK subgroup) also had PK analyses performed with a single dose of 50 IU/kg Advate (Advate Day 0) within 8 weeks prior to rFVIIIFc Day 0. A >= 96 hour washout was performed before the PK dose of Advate or rFVIIIFc was administered. Repeat PK profiling with a single dose of 50 IU/kg rFVIIIFc was conducted at Week 14 or after 12 to 24 weeks of prophylaxis with rFVIIIFc.
  After PK assessments, all participants started twice weekly treatment with 25 IU/kg of rFVIIIFc via intravenous (IV) injection on Day 1 and 50 IU/kg on Day 4, followed by individualized dose and interval modification within the range of 25 to 65 IU/kg every 3 to 5 days, as determined by rFVIIIFc PK analysis, to maintain a trough level of 1% to 3% (or higher, as clinically indicated) FVIII activity.
- Arm 2: Weekly Prophylaxis: 65 IU/kg of rFVIIIFc via IV injection every 7 days
- Arm 3: Episodic (On-Demand) Dosing: 10 to 50 IU/kg rFVIIIFc via IV injection, as required to treat a bleeding episode
Period: Overall Study
Arm/Group | Arm 1: Individualized (Tailored) Prophylaxis | Arm 2: Weekly Prophylaxis | Arm 3: Episodic (On-Demand) Dosing
Started | 118 | 24 | 23
Pharmacokinetic (PK) Subgroup | 30 | 0 | 0
Perioperative Management Subgroup | 8 (Participants who underwent major surgery.) | 1 (Participants who underwent major surgery.) | 0 (Participants who underwent major surgery.)
Completed | 112 | 19 | 22
Not Completed | 6 | 5 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Other | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Individualized (Tailored) Prophylaxis | Arm 2: Weekly Prophylaxis | Arm 3: Episodic (On-Demand) Dosing | Total
Number analyzed (Participants) | 118 | 24 | 23 | 165
Age, Continuous [Median (Full Range); unit: years] | 29.0 [12 to 65] | 31.5 [18 to 59] | 34.0 [13 to 62] | 30.0 [12 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 118 | 24 | 23 | 165

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of FVIII Inhibitor Development
Description: An inhibitor test result ≥0.6 Bethesda units (BU)/mL, identified and confirmed by re-testing of a second sample obtained within 2 to 4 weeks, was considered positive. Both tests were to be performed using the Nijmegen-modified Bethesda Assay by the central laboratory. The incidence rates along with the 95% confidence interval (CI) were summarized for all titers for subjects with 50 or more exposure days (EDs) to rFVIIIFc and a valid inhibitor test after the 50th exposure. In addition, the incidence rates for all subjects regardless of their exposure days to rFVIIIFc were also summarized. The 95% CI was calculated using Clopper-Pearson exact method.
Time Frame: up to 52 weeks ± 2 weeks
Population: Safety Analysis Set: participants who received at least 1 dose of Advate or at least 1 dose of rFVIIIFc; n=number of participants with given number of exposure days who had a valid inhibitor test.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- All Arms: Total: All participants from the Individualized (Tailored) Prophylaxis, Weekly Prophylaxis, and Episodic (On-Demand) Dosing arms.
Arm/Group | Arm 1: Individualized (Tailored) Prophylaxis | Arm 2: Weekly Prophylaxis | Arm 3: Episodic (On-Demand) Dosing | All Arms: Total
Number analyzed (Participants) | 118 | 24 | 23 | 165
percentage of participants
  Participants with>=50 EDs; n=107, 1, 2, 110 | 0 [0.0 to 3.4] | 0 [0.0 to 97.5] | 0 [0.0 to 84.2] | 0 [0.0 to 3.3]
  All participants; n=117, 24, 23, 164 | 0 [0.0 to 3.1] | 0 [0.0 to 14.2] | 0 [0.0 to 14.8] | 0 [0.0 to 2.2]

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: AE=any untoward medical occurrence that did not necessarily have a causal relationship with treatment, and could be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study product, whether related or not. TEAE=AE present prior to receiving the first injection of Advate or rFVIIIFc that subsequently worsened in severity or not present prior to receiving the first injection but subsequently appeared before the last visit on study. Serious AE (SAE)=AE resulting in death, immediate risk of death, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, or a congenital anomaly/birth defect, or any other medically important event. AEs emergent between the first Advate injection and first on-study rFVIIIFc injection (Sequential PK Subgroup) or during the surgical/rehabilitation period (Surgery Subgroup) are presented separately.
Time Frame: up to 52 weeks + 30 days ± 1 week
Population: Safety Analysis Set: participants who received at least 1 dose of Advate or at least 1 dose of rFVIIIFc. For Arm 1, AEs emergent between 1st on-study Advate dose and 1st rFVIIIFc dose are reported as treatment-emergent to Advate (1st column); AEs emergent after 1st rFVIIIFc injection are reported as treatment-emergent to rFVIIIFc (2nd column).
Measure: Number; unit: participants
Groups:
- Arm 1: Individualized (Tailored) Prophylaxis, Advate: Participants underwent pharmacokinetic (PK) analyses performed with a single dose of 50 IU/kg Advate (Advate Day 0) and then a single dose of 50 IU/kg rFVIIIFc (rFVIIIFc Day 0) within 8 weeks of the Advate dose. A >= 96 hour washout from Advate or any other FVIII product was performed before the PK dose of Advate or rFVIIIFc was administered. Repeat PK profiling with a single dose of 50 IU/kg rFVIIIFc was conducted at Week 14 or after 12 to 24 weeks of prophylaxis with rFVIIIFc.
  After PK assessments, participants started twice weekly treatment with 25 IU/kg of rFVIIIFc via IV injection on Day 1 and 50 IU/kg on Day 4, followed by individualized dose and interval modification within the range of 25 to 65 IU/kg every 3 to 5 days, as determined by rFVIIIFc PK analysis, to maintain a trough level of 1% to 3% (or higher, as clinically indicated) FVIII activity.
- Arm 1: Individualized (Tailored) Prophylaxis, rFVIIIFc Only: On rFVIIIFc Day 0, participants underwent pharmacokinetic (PK) analysis with a single dose of 50 IU/kg rFVIIIFc in order to estimate their PK parameters and guide the appropriate dose or interval of dosing.
  After the PK assessment, participants started twice weekly treatment with 25 IU/kg of rFVIIIFc via intravenous (IV) injection on Day 1 and 50 IU/kg on Day 4, followed by individualized dose and interval modification within the range of 25 to 65 IU/kg every 3 to 5 days, as determined by PK analyses, to maintain a trough level of 1% to 3% (or higher, as clinically indicated) FVIII activity.
- Any Arm: Perioperative Management (Surgery) Subgroup: Participants from any arm who underwent major surgery. The surgical period and dosing were dependent on the type of surgery the participant underwent.
Arm/Group | Arm 1: Individualized (Tailored) Prophylaxis, Advate | Arm 1: Individualized (Tailored) Prophylaxis, rFVIIIFc Only | Arm 2: Weekly Prophylaxis | Arm 3: Episodic (On-Demand) Dosing | Any Arm: Perioperative Management (Surgery) Subgroup
Number analyzed (Participants) | 30 | 117 | 24 | 23 | 9
participants
  >=1 TEAE | 3 | 80 | 18 | 10 | 4
  >=1 Related TEAE | 0 | 5 | 3 | 2 | 0
  >=1 TESAE | 0 | 10 | 2 | 0 | 2
  >=1 Related TESAE | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormal Laboratory Values From Baseline
Description: Clinical laboratory evaluations included hematology and blood chemistry. Table does not include laboratory tests evaluated during the surgical/rehabilitation period. ULN=upper limit of normal.
Time Frame: up to 52 weeks ± 2 weeks
Population: Safety Analysis Set: participants who received at least 1 dose of Advate or at least 1 dose of rFVIIIFc n=the number of participants with at least one post-baseline value.
Measure: Number; unit: participants
Arm/Group | Arm 1: Individualized (Tailored) Prophylaxis | Arm 2: Weekly Prophylaxis | Arm 3: Episodic (On-Demand) Dosing
Number analyzed (Participants) | 118 | 24 | 23
participants
  Leukocytes <3.0*10^9/L; n=117, 24, 23 | 2 | 0 | 2
  Leukocytes >=16*10^9/L; n=117, 24, 23 | 1 | 0 | 0
  Lymphocytes <0.8*10^9/L; n=104, 22, 21 | 3 | 1 | 1
  Lymphocytes >12*10^9/L; n=104, 22, 21 | 0 | 0 | 0
  Neutrophils <1.5*10^9/L; n=104, 22, 21 | 4 | 0 | 1
  Neutrophils >13.5*10^9/L; n=104, 22, 21 | 1 | 0 | 0
  Monocytes >2.5*10^9/L; n=104, 22, 21 | 0 | 0 | 0
  Eosinophils >1.6*10^9/L; n=104, 22, 21 | 0 | 0 | 0
  Basophils >1.6*10^9/L; n=104, 22, 21 | 0 | 0 | 0
  Erythrocytes <=3.5*10^12/L; n=117, 24, 23 | 1 | 0 | 0
  Erythrocytes >=6.4*10^12/L; n=117, 24, 23 | 1 | 0 | 1
  Hemoglobin <=115 g/L; n=117, 24, 23 | 3 | 0 | 1
  Hemoglobin >=190 g/L; n=117, 24, 23 | 0 | 0 | 0
  Hematocrit <=37%; n=117, 24, 23 | 5 | 2 | 1
  Hematocrit >=60%; n=117, 24, 23 | 0 | 0 | 0
  Platelets <=75*10^9/L; n=117, 24, 23 | 0 | 0 | 0
  Platelets >=700*10^9/L; n=117, 24, 23 | 0 | 0 | 0
  Alanine Aminotransferase >=3*ULN; n=117, 24, 23 | 4 | 0 | 0
  Aspartate Aminotransferase >=3*ULN; n=117, 24, 23 | 4 | 1 | 0
  Alkaline Phosphatase >=3*ULN; n=117, 24, 23 | 0 | 0 | 0
  Total Bilirubin >=34.2 µmol/L; n=117, 24, 23 | 3 | 0 | 2
  Blood Urea Nitrogen >=10.7 mmol/L; n=117, 24, 23 | 1 | 1 | 0
  Creatinine >=176.8 µmol/L; n=117, 24, 23 | 0 | 0 | 0
  Sodium <=126 mmol/L; n=117, 24, 23 | 0 | 0 | 0
  Sodium >=156 mmol/L; n=117, 24, 23 | 1 | 0 | 0
  Potassium <=3 mmol/L; n=117, 24, 23 | 0 | 0 | 0
  Potassium >=6 mmol/L; n=117, 24, 23 | 0 | 0 | 0
  Chloride <=90 mmol/L; n=117, 24, 23 | 1 | 0 | 0
  Chloride >=118 mmol/L; n=117, 24, 23 | 0 | 0 | 0
  Phosphate <=0.55 mmol/L n=117, 24, 23 | 1 | 0 | 0
  Phosphate >=1.71 mmol/L; n=117, 24, 23 | 0 | 0 | 0
  Glucose <=2.22 mmol/L; n=117, 24, 23 | 0 | 0 | 0
  Glucose >=9.71 mmol/L; n=117, 24, 23 | 2 | 1 | 0
  Total Protein <=45 g/L; n=117, 24, 23 | 0 | 0 | 0
  Total Protein >=100 g/L; n=117, 24, 23 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Relevant Abnormalities in Vital Signs or Relevant Changes From Baseline in Vital Signs
Description: Number of participants with clinically relevant abnormalities or relevant changes from baseline in temperature, pulse (beats per minute [bpm]), systolic blood pressure (SBP), and diastolic blood pressure (DBP) are presented. Baseline (BL) is defined as the last non-missing evaluable assessment taken prior and closest to the first rFVIIIFc dose. ↑ signifies increase and ↓ signifies decrease.
Time Frame: up to 52 weeks ± 2 weeks
Population: Safety Analysis Set: participants who received at least 1 dose of Advate or at least 1 dose of rFVIIIFc and had a baseline assessment and at least one post-baseline assessment for temperature or at least one post-baseline assessment for pulse, systolic blood pressure, and diastolic blood pressure.
Measure: Number; unit: participants
Arm/Group | Arm 1: Individualized (Tailored) Prophylaxis | Arm 2: Weekly Prophylaxis | Arm 3: Episodic (On-Demand) Dosing
Number analyzed (Participants) | 113 | 24 | 23
participants
  Temperature: >38°C and ≥1°C ↑ from BL | 1 | 0 | 0
  Pulse: >120 bpm or >20 bpm ↑ from BL | 11 | 2 | 0
  Pulse: <50 bpm or >20 bpm ↓ from BL | 11 | 2 | 1
  SBP: >180 mm Hg or >40 mm Hg ↑ from BL | 0 | 1 | 0
  SBP: <90 mm Hg or >30 mm Hg ↓ from BL | 5 | 1 | 1
  DBP: >105 mm Hg or >30 mm Hg ↑ from BL | 1 | 0 | 0
  DBP: <50 mm Hg or >20 mm Hg ↓ from BL | 5 | 0 | 1

5. Primary Outcome: Annualized Bleeding Rate
Description: Annualized bleeding episodes = (number of bleeding episodes during the efficacy period / number of days during the efficacy period)*365.25. The efficacy period in Arms 1 and 2 began with the first prophylactic dose of rFVIIIFc and ended with the last dose (regardless of reason for dosing). The efficacy period in Arm 3 began at the time of last PK rFVIIIFc sampling timepoint and ended at the date of the last study visit. Periods of PK evaluations and surgery/rehabilitation are not included in the efficacy period. A bleeding episode started from the first sign of a bleed, and ended 72 hours after the last treatment for the bleeding, within which any symptoms of bleeding at the same location, or injections less than or equal to 72 hours apart, were considered the same bleeding episode.
Time Frame: up to 52 weeks ± 2 weeks (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFVIIIFc with an efficacy assessment.
Measure: Median (Inter-Quartile Range); unit: episodes per participant per year
Arm/Group | Arm 1: Individualized (Tailored) Prophylaxis | Arm 2: Weekly Prophylaxis | Arm 3: Episodic (On-Demand) Dosing
Number analyzed (Participants) | 117 | 23 | 23
episodes per participant per year | 1.60 [0.00 to 4.69] | 3.59 [1.86 to 8.36] | 33.57 [21.14 to 48.69]

6. Primary Outcome: Comparison of Annualized Bleeding Rates: Arm 1 Versus Arm 3
Description: Estimated using the negative binomial model with treatment arm as covariate, based on whole study duration for all participants. Annualized bleeding episodes = (number of bleeding episodes / number of days in the respective period)*365.25.The efficacy period in Arm 1 began with the first prophylactic dose of rFVIIIFc and ended with the last dose (regardless of reason for dosing). The efficacy period in Arm 3 began at the time of last PK rFVIIIFc sampling timepoint and ended at the date of the last study visit. Periods of PK evaluations and surgery/rehabilitation are not included in the efficacy period. A bleeding episode started from the first sign of a bleed, and ended 72 hours after the last treatment for the bleeding, within which any symptoms of bleeding at the same location, or injections less than or equal to 72 hours apart, were considered part of the same bleeding episode.
Time Frame: up to 52 weeks ± 2 weeks (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFVIIIFc with an efficacy assessment.
Measure: Number (95% Confidence Interval); unit: episodes per participant per year
Arm/Group | Arm 1: Individualized (Tailored) Prophylaxis | Arm 3: Episodic (On-Demand) Dosing
Number analyzed (Participants) | 117 | 23
episodes per participant per year | 2.91 [2.30 to 3.68] | 37.25 [24.03 to 57.74]
Statistical Analysis 1: Comparison: Arm 1: Individualized (Tailored) Prophylaxis vs Arm 3: Episodic (On-Demand) Dosing; The null hypothesis for the primary endpoint is no difference between the individualized (tailored) prophylaxis regimen and the on-demand regimen. The sample size of this study was mainly based on clinical rather than statistical considerations. However it was projected to have > 90% power at the 2-sided 0.05 level of significance to detect a 60% reduction in annualized bleeding episodes, based upon this hypothesis test; Test type: Superiority or Other; p < 0.001, negative binomial model; Bleeding Rate Ratio = 0.08, 95% CI 2-sided [0.05 to 0.13]

7. Primary Outcome: Area Under the Curve (AUC) Per Dose (One-stage Clotting Assay)
Description: Dose normalized area under the drug concentration-time curve. Sampling for Advate PK profiling was conducted, following at least 96 hours of washout, at these timepoints: preinjection and at either 30 (±3) minutes or 10 (±3) minutes, 1 hour (±15 minutes), 6 (±1) hours, 24 (±2) hours (Day 1), 48 (±2) hours (Day 2), and 72 (±2) hours (Day 3) from the start of the injection. Sampling for rFVIIIFc PK profiling was conducted at Day 0 (directly following at least 96 hours washout from Advate PK profiling or within 4 weeks of the Advate dose or other rFVIII product) and repeated 12 to 24 weeks later at the following timepoints: preinjection and at 30 (±3) minutes (or 10 (±3) minutes), 1 hour (±15 minutes), 6 (±1) hours, 24 (±2) hours (Day 1), 72 (±2) hours (Day 3), 96 (±2) hours (Day 4), and 120 (±2) hours (Day 5) from the start of the injection.
Time Frame: See Measure Description for complete time frame.
Population: Participants who had evaluable one-stage PK profiles for both Advate and baseline rFVIIIFc.
Measure: Geometric Mean (95% Confidence Interval); unit: IU*h/dL per IU/kg
Groups:
- Individualized (Tailored) Prophylaxis: Sequential PK Subgroup: On rFVIIIFc Day 0, all participants underwent pharmacokinetic (PK) analysis with 50 IU/kg rFVIIIFc to estimate their PK parameters and guide the appropriate dose or interval of dosing. A subset of participants (Sequential PK subgroup) also had PK analyses performed with a single dose of 50 IU/kg Advate (Advate Day 0) within 8 weeks prior to rFVIIIFc Day 0. A >= 96 hour washout was performed before the PK dose of Advate or rFVIIIFc was administered. Repeat PK profiling with a single dose of 50 IU/kg rFVIIIFc was conducted at Week 14 or after 12 to 24 weeks of prophylaxis with rFVIIIFc.
  After PK assessments, all participants started twice weekly treatment with 25 IU/kg of rFVIIIFc via intravenous (IV) injection on Day 1 and 50 IU/kg on Day 4, followed by individualized dose and interval modification within the range of 25 to 65 IU/kg every 3 to 5 days, as determined by rFVIIIFc PK analysis, to maintain a trough level of 1% to 3% (or higher, as clinically indicated) FVIII activity.
Arm/Group | Individualized (Tailored) Prophylaxis: Sequential PK Subgroup
Number analyzed (Participants) | 28
IU*h/dL per IU/kg
  rFVIIIFc Baseline | 51.24 [44.97 to 58.38]
  Advate | 32.88 [29.31 to 36.88]

8. Primary Outcome: Elimination Half Life (t1/2; One-stage Clotting Assay)
Description: Time required for the activity of the drug to reach half of its original value. Sampling for Advate PK profiling was conducted, following at least 96 hours of washout, at these timepoints: preinjection and at either 30 (±3) minutes or 10 (±3) minutes, 1 hour (±15 minutes), 6 (±1) hours, 24 (±2) hours (Day 1), 48 (±2) hours (Day 2), and 72 (±2) hours (Day 3) from the start of the injection. Sampling for rFVIIIFc PK profiling was conducted at Day 0 (directly following at least 96 hours washout from Advate PK profiling or within 4 weeks of the Advate dose or other rFVIII product) and repeated 12 to 24 weeks later at the following timepoints: preinjection and at 30 (±3) minutes (or 10 (±3) minutes), 1 hour (±15 minutes), 6 (±1) hours, 24 (±2) hours (Day 1), 72 (±2) hours (Day 3), 96 (±2) hours (Day 4), and 120 (±2) hours (Day 5) from the start of the injection.
Time Frame: See Measure Description for complete time frame.
Population: Participants who had evaluable one-stage PK profiles for both Advate and baseline rFVIIIFc.
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Individualized (Tailored) Prophylaxis: Sequential PK Subgroup
Number analyzed (Participants) | 28
hours
  rFVIIIFc Baseline | 18.97 [17.03 to 21.12]
  Advate | 12.43 [11.14 to 13.86]

9. Primary Outcome: Clearance (CL; One-stage Clotting Assay)
Description: Rate at which the body removes the drug, measured as the volume of the plasma cleared of drug per unit time per unit weight. Sampling for Advate PK profiling was conducted, following at least 96 hours of washout, at these timepoints: preinjection and at either 30 (±3) minutes or 10 (±3) minutes, 1 hour (±15 minutes), 6 (±1) hours, 24 (±2) hours (Day 1), 48 (±2) hours (Day 2), and 72 (±2) hours (Day 3) from the start of the injection. Sampling for rFVIIIFc PK profiling was conducted at Day 0 (directly following at least 96 hours washout from Advate PK profiling or within 4 weeks of the Advate dose or other rFVIII product) and repeated 12 to 24 weeks later at the following timepoints: preinjection and at 30 (±3) minutes (or 10 (±3) minutes), 1 hour (±15 minutes), 6 (±1) hours, 24 (±2) hours (Day 1), 72 (±2) hours (Day 3), 96 (±2) hours (Day 4), and 120 (±2) hours (Day 5) from the start of the injection.
Time Frame: See Measure Description for complete time frame.
Population: Participants who had evaluable one-stage PK profiles for both Advate and baseline rFVIIIFc.
Measure: Geometric Mean (95% Confidence Interval); unit: mL/h/kg
Arm/Group | Individualized (Tailored) Prophylaxis: Sequential PK Subgroup
Number analyzed (Participants) | 28
mL/h/kg
  rFVIIIFc Baseline | 1.952 [1.713 to 2.224]
  Advate | 3.041 [2.711 to 3.412]

10. Primary Outcome: Mean Residence Time (MRT; One-stage Clotting Assay)
Description: The average time that a drug molecule is present in the systemic circulation. Sampling for Advate PK profiling was conducted, following at least 96 hours of washout, at these timepoints: preinjection and at either 30 (±3) minutes or 10 (±3) minutes, 1 hour (±15 minutes), 6 (±1) hours, 24 (±2) hours (Day 1), 48 (±2) hours (Day 2), and 72 (±2) hours (Day 3) from the start of the injection. Sampling for rFVIIIFc PK profiling was conducted at Day 0 (directly following at least 96 hours washout from Advate PK profiling or within 4 weeks of the Advate dose or other rFVIII product) and repeated 12 to 24 weeks later at the following timepoints: preinjection and at 30 (±3) minutes (or 10 (±3) minutes), 1 hour (±15 minutes), 6 (±1) hours, 24 (±2) hours (Day 1), 72 (±2) hours (Day 3), 96 (±2) hours (Day 4), and 120 (±2) hours (Day 5) from the start of the injection.
Time Frame: See Measure Description for complete time frame.
Population: Participants who had evaluable one-stage PK profiles for both Advate and baseline rFVIIIFc.
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Individualized (Tailored) Prophylaxis: Sequential PK Subgroup
Number analyzed (Participants) | 28
hours
  rFVIIIFc Baseline | 25.15 [22.65 to 27.91]
  Advate | 16.84 [15.22 to 18.63]

11. Primary Outcome: Incremental Recovery (One-stage Clotting Assay)
Description: The rise in FVIII activity in IU/dL per unit dose administered in IU/kg. Sampling for Advate PK profiling was conducted, following at least 96 hours of washout, at these timepoints: preinjection and at either 30 (±3) minutes or 10 (±3) minutes, 1 hour (±15 minutes), 6 (±1) hours, 24 (±2) hours (Day 1), 48 (±2) hours (Day 2), and 72 (±2) hours (Day 3) from the start of the injection. Sampling for rFVIIIFc PK profiling was conducted at Day 0 (directly following at least 96 hours washout from Advate PK profiling or within 4 weeks of the Advate dose or other rFVIII product) and repeated 12 to 24 weeks later at the following timepoints: preinjection and at 30 (±3) minutes (or 10 (±3) minutes), 1 hour (±15 minutes), 6 (±1) hours, 24 (±2) hours (Day 1), 72 (±2) hours (Day 3), 96 (±2) hours (Day 4), and 120 (±2) hours (Day 5) from the start of the injection.
Time Frame: See Measure Description for complete time frame.
Population: Participants who had evaluable one-stage PK profiles for both Advate and baseline rFVIIIFc.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL per IU/kg
Arm/Group | Individualized (Tailored) Prophylaxis: Sequential PK Subgroup
Number analyzed (Participants) | 28
IU/dL per IU/kg
  rFVIIIFc Baseline | 2.2395 [2.1116 to 2.3753]
  Advate | 2.3516 [2.2110 to 2.5010]

12. Secondary Outcome: Comparison of Annualized Bleeding Rates: Arm 2 Versus Arm 3
Description: Estimated using the negative binomial model with treatment arm as covariate, based on whole study duration for all participants. Annualized bleeding episodes = (number of bleeding episodes / number of days in the respective period)*365.25.The efficacy period in Arm 2 began with the first prophylactic dose of rFVIIIFc and ended with the last dose (regardless of reason for dosing). The efficacy period in Arm 3 began at the time of last PK rFVIIIFc sampling timepoint and ended at the date of the last study visit. Periods of PK evaluations and surgery/rehabilitation are not included in the efficacy period. A bleeding episode started from the first sign of a bleed, and ended 72 hours after the last treatment for the bleeding, within which any symptoms of bleeding at the same location, or injections less than or equal to 72 hours apart, were considered the same bleeding episode.
Time Frame: up to 52 weeks ± 2 weeks (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFVIIIFc with an efficacy assessment.
Measure: Number (95% Confidence Interval); unit: episodes per participant per year
Arm/Group | Arm 2: Weekly Prophylaxis | Arm 3: Episodic (On-Demand) Dosing
Number analyzed (Participants) | 23 | 23
episodes per participant per year | 8.92 [5.48 to 14.51] | 37.25 [24.03 to 57.74]
Statistical Analysis 1: Comparison: Arm 2: Weekly Prophylaxis vs Arm 3: Episodic (On-Demand) Dosing; Test type: Superiority or Other; p < 0.001, negative binomial model; Bleeding Rate Ratio = 0.24, 95% CI 2-sided [0.12 to 0.46]

13. Secondary Outcome: Annualized rFVIIIFc Consumption Per Participant
Description: Consumption is calculated for the efficacy period. The efficacy period in Arms 1 and 2 began with the first prophylactic dose of rFVIIIFc and ended with the last dose (regardless of reason for dosing). The efficacy period in Arm 3 began at the time of last PK rFVIIIFc sampling timepoint and ended at the date of the last study visit. Periods of PK evaluations and surgery/rehabilitation are not included in the efficacy period. Overall units (IU/kg) of annualized rFVIIIFc consumption = [Total rFVIIIFc IU/kg received during the efficacy period / number of days in efficacy period] x 365.25.
Time Frame: up to 52 weeks ± 2 weeks (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFVIIIFc. 'Overall' n=participants in the Full Analysis Set with evaluable data in the efficacy period; 'Last 3 Months on Study' n=participants in the Full Analysis Set with evaluable data and >=6 months on study.
Measure: Mean (Standard Deviation); unit: IU/kg rFVIIIFc per participant per year
Arm/Group | Arm 1: Individualized (Tailored) Prophylaxis | Arm 2: Weekly Prophylaxis | Arm 3: Episodic (On-Demand) Dosing
Number analyzed (Participants) | 117 | 24 | 23
IU/kg rFVIIIFc per participant per year
  Overall (n=117, 23, 23) | 4631.98 (1041.608) | 4003.69 (652.573) | 1304.36 (874.361)
  Last 3 months on study (n=112, 16, 18) | 4868.35 (1365.108) | 3882.89 (583.344) | 1225.80 (848.656)

14. Secondary Outcome: Participant Assessment of Response to Injections to Treat a Bleeding Episode
Description: Participant's assessment of the response to the first rFVIIIFc injection for each bleeding episode. Percentages were based on the number of bleeding episodes for which a response was provided for the first injection, using the following 4-point scale: excellent=abrupt pain relief and/or improvement in signs of bleeding within approximately 8 hours after the initial injection; good=definite pain relief and/or improvement in signs of bleeding within approximately 8 hours after an injection, but possibly requiring more than one injection after 24 to 48 hours for complete resolution; moderate=probable or slight beneficial effect within 8 hours after the initial injection and requiring more than one injection; no response=no improvement, or condition worsened, within approximately 8 hours after the initial injection.
Time Frame: up to 52 weeks ± 2 weeks
Population: Full Analysis Set: participants who received at least 1 dose of rFVIIIFc and had at least 1 evaluable bleeding episode; based on the number of injections with an evaluation.
Measure: Number; unit: percentage of responses
Units Other Than Participants: Bleeding Episodes
Arm/Group | Arm 1: Individualized (Tailored) Prophylaxis | Arm 2: Weekly Prophylaxis | Arm 3: Episodic (On-Demand) Dosing
Number analyzed (Participants) | 63 | 19 | 23
Number analyzed (Bleeding Episodes) | 202 | 89 | 454
percentage of responses
  Excellent or Good | 79.7 | 64.0 | 80.2
  Excellent | 33.7 | 18.0 | 30.8
  Good | 46.0 | 46.1 | 49.3
  Moderate | 18.8 | 34.8 | 19.6
  No Response | 1.5 | 1.1 | 0.2

15. Secondary Outcome: Investigator's Assessment of Participants' Bleeding Response to rFVIIIFc Injection
Description: The investigator was given the opportunity to record an assessment of a participant's response to treatment, if the participant was treated in the hospital for a major bleed, using the following 4-point scale: excellent=abrupt pain relief and/or improvement in signs of bleeding within approximately 8 hours after the initial injection; good=definite pain relief and/or improvement in signs of bleeding within approximately 8 hours after an injection, but possibly requiring more than one injection after 24 to 48 hours for complete resolution; moderate=probable or slight beneficial effect within 8 hours after the initial injection and requiring more than one injection; no response=no improvement, or condition worsened, within approximately 8 hours after the initial injection.
Time Frame: up to 52 weeks ± 2 weeks
Population: This supplemental assessment was not summarized because of insufficient data.
Arm/Group | Arm 1: Individualized (Tailored) Prophylaxis | Arm 2: Weekly Prophylaxis | Arm 3: Episodic (On-Demand) Dosing
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Annualized Bleeding Rate by Location of Bleed (Joint, Muscle, Internal, Skin/Mucosa)
Description: Annualized bleeding episodes = (Number of bleeding episodes at the specified location / number of days in efficacy period) x 365.25. The efficacy period in Arms 1 and 2 began with the first prophylactic dose of rFVIIIFc and ended with the last dose (regardless of reason for dosing). The efficacy period in Arm 3 began at the time of last PK rFVIIIFc sampling timepoint and ended at the date of the last study visit. Periods of PK evaluations and surgery/rehabilitation were not included in the efficacy period. A bleeding episode started from the first sign of a bleed, and ended 72 hours after the last treatment for the bleeding, within which any symptoms of bleeding at the same location, or injections less than or equal to 72 hours apart, were considered the same bleeding episode. Any bleeding at a different location was a separate bleeding episode regardless of time from the last injection.
Time Frame: up to 52 weeks ± 2 weeks (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFVIIIFc with evaluable data.
Measure: Median (Inter-Quartile Range); unit: episodes per participant per year
Arm/Group | Arm 1: Individualized (Tailored) Prophylaxis | Arm 2: Weekly Prophylaxis | Arm 3: Episodic (On-Demand) Dosing
Number analyzed (Participants) | 117 | 23 | 23
episodes per participant per year
  Joint | 0.00 [0.00 to 3.11] | 1.93 [0.00 to 7.62] | 22.76 [15.07 to 39.02]
  Muscle | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 2.01] | 5.57 [1.86 to 10.05]
  Internal | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Soft Tissue | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 1.86]
  Skin/Mucosa | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

17. Secondary Outcome: Annualized Joint Bleeding Rate (Spontaneous and Traumatic)
Description: Annualized bleeding episodes = (Number of bleeding episodes of the specified type / number of days in efficacy period) x 365.25. The efficacy period in Arms 1 and 2 began with the first prophylactic dose of rFVIIIFc and ended with the last dose (regardless of reason for dosing). The efficacy period in Arm 3 began at the time of last PK rFVIIIFc sampling timepoint and ended at the date of the last study visit. Periods of PK evaluations and surgery/rehabilitation were not included in the efficacy period. A bleeding episode started from the first sign of a bleed, and ended 72 hours after the last treatment for the bleeding, within which any symptoms of bleeding at the same location, or injections less than or equal to 72 hours apart, were considered the same bleeding episode.
Time Frame: up to 52 weeks ± 2 weeks (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFVIIIFc with evaluable data.
Measure: Median (Inter-Quartile Range); unit: bleeding episodes per participant per yr
Arm/Group | Arm 1: Individualized (Tailored) Prophylaxis | Arm 2: Weekly Prophylaxis | Arm 3: Episodic (On-Demand) Dosing
Number analyzed (Participants) | 117 | 23 | 23
bleeding episodes per participant per yr
  Spontaneous | 0.00 [0.00 to 1.73] | 0.00 [0.00 to 3.81] | 18.59 [7.59 to 29.59]
  Traumatic | 0.00 [0.00 to 1.16] | 0.00 [0.00 to 2.01] | 3.93 [0.00 to 8.56]
  Unknown | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

18. Secondary Outcome: Number of Days From Last Treatment Injection to a New Bleeding Episode
Description: Number of days from the last injection to treat a bleeding episode to a new bleeding episode, analyzed for per evaluable bleeding episode and per participant. For "per participant" values, number of days from last injection to treat a bleed to a new bleeding episode is averaged across all evaluable bleeding episodes for each participant first, and then descriptive statistics were calculated across participants. A follow-up injection administered >72 hours after the most recent injection given to treat a bleed was considered a new bleed at the same location and was classified as type=Unknown (not evaluable). The efficacy period in Arms 1 and 2 began with the first prophylactic dose of rFVIIIFc and ended with the last dose (regardless of reason for dosing). The efficacy period in Arm 3 began at the time of last PK rFVIIIFc sampling timepoint and ended at the date of the last study visit. Periods of PK evaluations and surgery/rehabilitation were not included in the efficacy period.
Time Frame: up to 52 weeks ± 2 weeks (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFVIIIFc and had at least 1 evaluable bleeding episode. The first bleed for each participant could not be included in this analysis since there was no previous bleed from which to measure time.
Measure: Median (Inter-Quartile Range); unit: days
Units Other Than Participants: Evaluable Bleeding Episodes
Arm/Group | Arm 1: Individualized (Tailored) Prophylaxis | Arm 2: Weekly Prophylaxis | Arm 3: Episodic (On-Demand) Dosing
Number analyzed (Participants) | 48 | 12 | 23
Number analyzed (Evaluable Bleeding Episodes) | 149 | 76 | 430
days
  Per Bleeding Episode | 19.83 [8.58 to 55.46] | 8.00 [5.35 to 15.38] | 6.55 [4.46 to 10.27]
  Per Participant | 42.90 [20.25 to 65.93] | 40.71 [11.75 to 52.39] | 10.12 [7.42 to 16.37]

19. Secondary Outcome: Number of Injections Required for Resolution of a Bleeding Episode
Description: A bleeding episode started from the first sign of a bleed, and ended 72 hours after the last treatment for the bleeding, within which any symptoms of bleeding at the same location, or injections less than or equal to 72 hours apart, were considered the same bleeding episode. All injections given from the initial sign of a bleed until the last date/time within the bleed window are counted. The resolution of a bleed is defined as no sign of bleeding following injection for the bleed. The efficacy period in Arms 1 and 2 began with the first prophylactic dose of rFVIIIFc and ended with the last dose (regardless of reason for dosing). The efficacy period in Arm 3 began at the time of last PK rFVIIIFc sampling timepoint and ended at the date of the last study visit. Periods of PK evaluations and surgery/rehabilitation are not included in the efficacy period.
Time Frame: up to 52 weeks ± 2 weeks (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFVIIIFc and had at least 1 bleeding episode.
Measure: Median (Inter-Quartile Range); unit: injections
Units Other Than Participants: Bleeding Episodes
Arm/Group | Arm 1: Individualized (Tailored) Prophylaxis | Arm 2: Weekly Prophylaxis | Arm 3: Episodic (On-Demand) Dosing
Number analyzed (Participants) | 64 | 19 | 23
Number analyzed (Bleeding Episodes) | 209 | 92 | 456
injections
  Per Bleeding Episode | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Per Participant | 1.00 [1.00 to 1.33] | 1.00 [1.00 to 1.43] | 1.03 [1.00 to 1.17]

20. Secondary Outcome: Number of Injections Required for Resolution of a Bleeding Episode by Location of Bleed
Description: Please see Outcome Measure 20 for a definition of the efficacy period. A bleeding episode started from the first sign of a bleed, and ended 72 hours after the last treatment for the bleeding, within which any symptoms of bleeding at the same location, or injections less than or equal to 72 hours apart, were considered the same bleeding episode. All injections given from the initial sign of a bleed until the last date/time within the bleed window were counted. The resolution of a bleed was defined as no sign of bleeding following injection for the bleed. Bleeding episodes that presented in multiple locations are included as a single event in the overall summary for the number of injections to resolve that bleeding episode but are included in summaries for each location.
Time Frame: up to 52 weeks ± 2 weeks (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFVIIIFc and had evaluable efficacy assessments; n=total number of bleeds at given location.
Measure: Median (Inter-Quartile Range); unit: injections
Arm/Group | Arm 1: Individualized (Tailored) Prophylaxis | Arm 2: Weekly Prophylaxis | Arm 3: Episodic (On-Demand) Dosing
Number analyzed (Participants) | 64 | 19 | 23
injections
  Joint (n=151, 67, 366) | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Muscle (n=35, 23, 82) | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Soft Tissue (n=24, 5, 25) | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0]
  Internal (n=3, 2, 6) | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Skin/Mucosa (n=11, 6, 8) | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]

21. Secondary Outcome: Total Dose Per Injection Required for Resolution of a Bleeding Episode by Location of Bleed
Description: For each bleeding episode at one location, the total dose is the sum of the doses (IU/kg) administered across all injections given to treat that bleeding episode. Please see Outcome Measure 20 for a definition of the efficacy period. A bleeding episode started from the first sign of a bleed, and ended 72 hours after the last treatment for the bleeding, within which any symptoms of bleeding at the same location, or injections less than or equal to 72 hours apart, were considered part of the same bleeding episode. Bleeding episodes that presented in multiple locations are included as a single event in the overall summary for dose administered to resolve that bleeding episode but are included in the individual summaries for each location.
Time Frame: up to 52 weeks ± 2 weeks (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFVIIIFc and had complete information on the dose administered to treat a bleeding episode; n=total number of bleeding episodes at this location.
Measure: Median (Inter-Quartile Range); unit: IU/kg
Arm/Group | Arm 1: Individualized (Tailored) Prophylaxis | Arm 2: Weekly Prophylaxis | Arm 3: Episodic (On-Demand) Dosing
Number analyzed (Participants) | 63 | 19 | 23
IU/kg
  Joint (n=151, 67, 366) | 29.69 [24.10 to 53.44] | 28.23 [20.16 to 40.32] | 27.35 [22.73 to 39.22]
  Muscle (n=35, 23, 82) | 40.98 [26.79 to 53.10] | 32.12 [26.98 to 32.47] | 27.78 [23.47 to 31.01]
  Soft Tissue (n=23, 5, 25) | 30.60 [24.51 to 53.13] | 51.88 [20.16 to 54.88] | 27.78 [23.44 to 31.45]
  Internal (n=3, 2, 6) | 32.63 [23.39 to 51.72] | 58.40 [48.08 to 68.73] | 32.54 [30.00 to 49.18]
  Skin/Mucosa (n=11, 6, 8) | 33.90 [28.23 to 53.19] | 28.34 [21.65 to 44.35] | 21.37 [19.95 to 25.16]

22. Secondary Outcome: Volume at Steady State (Vss; One-stage Clotting Assay)
Description: Volume of distribution at steady state. Sampling for Advate PK profiling was conducted, following at least 96 hours of washout, at these timepoints: preinjection and at either 30 (±3) minutes or 10 (±3) minutes, 1 hour (±15 minutes), 6 (±1) hours, 24 (±2) hours (Day 1), 48 (±2) hours (Day 2), and 72 (±2) hours (Day 3) from the start of the injection. Sampling for rFVIIIFc PK profiling was conducted at Day 0 (directly following at least 96 hours washout from Advate PK profiling or within 4 weeks of the Advate dose or other rFVIII product) and repeated 12 to 24 weeks later at the following timepoints: preinjection and at 30 (±3) minutes (or 10 (±3) minutes), 1 hour (±15 minutes), 6 (±1) hours, 24 (±2) hours (Day 1), 72 (±2) hours (Day 3), 96 (±2) hours (Day 4), and 120 (±2) hours (Day 5) from the start of the injection.
Time Frame: See Measure Description for complete time frame.
Population: Participants who had evaluable one-stage PK profiles for both Advate and baseline rFVIIIFc.
Measure: Geometric Mean (95% Confidence Interval); unit: mL/kg
Arm/Group | Individualized (Tailored) Prophylaxis: Sequential PK Subgroup
Number analyzed (Participants) | 28
mL/kg
  rFVIIIFc Baseline | 49.1 [46.6 to 51.7]
  Advate | 51.2 [47.2 to 55.5]

23. Secondary Outcome: Volume at Steady State (Vss; Two-stage Chromogenic Assay)
Description: as for outcome 22
Time Frame: See Measure Description for complete time frame.
Population: Participants who had evaluable two-stage PK profiles for both Advate and baseline rFVIIIFc.
Measure: Geometric Mean (95% Confidence Interval); unit: mL/kg
Arm/Group | Individualized (Tailored) Prophylaxis: Sequential PK Subgroup
Number analyzed (Participants) | 27
mL/kg
  rFVIIIFc Baseline | 52.6 [47.4 to 58.3]
  Advate | 56.8 [51.5 to 62.7]

24. Secondary Outcome: Time to 1% and 3% FVIII Activity (One-stage Clotting Assay)
Description: Estimated time after dose (in days) when FVIII activity has declined to approximately 1 or 3 IU/dL (1% or 3%) above baseline, respectively. Sampling for Advate PK profiling was conducted, following at least 96 hours of washout, at these timepoints: preinjection and at either 30 (±3) minutes or 10 (±3) minutes, 1 hour (±15 minutes), 6 (±1) hours, 24 (±2) hours (Day 1), 48 (±2) hours (Day 2), and 72 (±2) hours (Day 3) from the start of the injection. Sampling for rFVIIIFc PK profiling was conducted at Day 0 (directly following at least 96 hours washout from Advate PK profiling or within 4 weeks of the Advate dose or other rFVIII product) and repeated 12 to 24 weeks later at the following timepoints: preinjection and at 30 (±3) minutes (or 10 (±3) minutes), 1 hour (±15 minutes), 6 (±1) hours, 24 (±2) hours (Day 1), 72 (±2) hours (Day 3), 96 (±2) hours (Day 4), and 120 (±2) hours (Day 5) from the start of the injection.
Time Frame: See Measure Description for complete time frame.
Population: Participants who had evaluable one-stage PK profiles for both Advate and baseline rFVIIIFc.
Measure: Geometric Mean (95% Confidence Interval); unit: days
Arm/Group | Individualized (Tailored) Prophylaxis: Sequential PK Subgroup
Number analyzed (Participants) | 28
days
  Advate: Time 1% | 3.298 [2.985 to 3.645]
  Advate: Time 3% | 2.478 [2.242 to 2.738]
  rFVIIIFc Baseline: Time 1% | 4.918 [4.434 to 5.455]
  rFVIIIFc Baseline: Time 3% | 3.707 [3.325 to 4.133]

25. Secondary Outcome: Time to 1% and 3% FVIII Activity (Two-stage Chromogenic Assay)
Description: as for outcome 24
Time Frame: See Measure Description for complete time frame.
Population: Participants who had evaluable two-stage PK profiles for both Advate and baseline rFVIIIFc.
Measure: Geometric Mean (95% Confidence Interval); unit: days
Arm/Group | Individualized (Tailored) Prophylaxis: Sequential PK Subgroup
Number analyzed (Participants) | 27
days
  Advate: Time 1% | 3.220 [2.970 to 3.491]
  Advate: Time 3% | 2.306 [2.120 to 2.509]
  rFVIIIFc Baseline: Time 1% | 5.010 [4.525 to 5.548]
  rFVIIIFc Baseline: Time 3% | 3.612 [3.250 to 4.015]

26. Secondary Outcome: Time at Maximum Activity (Tmax; One-stage Clotting Assay)
Description: Time at which maximum activity (Cmax) is observed. Sampling for Advate PK profiling was conducted, following at least 96 hours of washout, at these timepoints: preinjection and at either 30 (±3) minutes or 10 (±3) minutes, 1 hour (±15 minutes), 6 (±1) hours, 24 (±2) hours (Day 1), 48 (±2) hours (Day 2), and 72 (±2) hours (Day 3) from the start of the injection. Sampling for rFVIIIFc PK profiling was conducted at Day 0 (directly following at least 96 hours washout from Advate PK profiling or within 4 weeks of the Advate dose or other rFVIII product) and repeated 12 to 24 weeks later at the following timepoints: preinjection and at 30 (±3) minutes (or 10 (±3) minutes), 1 hour (±15 minutes), 6 (±1) hours, 24 (±2) hours (Day 1), 72 (±2) hours (Day 3), 96 (±2) hours (Day 4), and 120 (±2) hours (Day 5) from the start of the injection.
Time Frame: See Measure Description for complete time frame.
Population: Participants who had evaluable one-stage PK profiles for both Advate and baseline rFVIIIFc.
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Individualized (Tailored) Prophylaxis: Sequential PK Subgroup
Number analyzed (Participants) | 28
hours
  rFVIIIFc Baseline | 0.49 [0.37 to 0.63]
  Advate | 0.48 [0.33 to 0.68]

27. Secondary Outcome: Time at Maximum Activity (Tmax; Two-stage Chromogenic Assay)
Description: Time at which the maximum activity (Cmax) is observed. Sampling for Advate PK profiling was conducted, following at least 96 hours of washout, at these timepoints: preinjection and at either 30 (±3) minutes or 10 (±3) minutes, 1 hour (±15 minutes), 6 (±1) hours, 24 (±2) hours (Day 1), 48 (±2) hours (Day 2), and 72 (±2) hours (Day 3) from the start of the injection. Sampling for rFVIIIFc PK profiling was conducted at Day 0 (directly following at least 96 hours washout from Advate PK profiling or within 4 weeks of the Advate dose or other rFVIII product) and repeated 12 to 24 weeks later at the following timepoints: preinjection and at 30 (±3) minutes (or 10 (±3) minutes), 1 hour (±15 minutes), 6 (±1) hours, 24 (±2) hours (Day 1), 72 (±2) hours (Day 3), 96 (±2) hours (Day 4), and 120 (±2) hours (Day 5) from the start of the injection.
Time Frame: See Measure Description for complete time frame.
Population: Participants who had evaluable two-stage PK profiles for both Advate and baseline rFVIIIFc.
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Individualized (Tailored) Prophylaxis: Sequential PK Subgroup
Number analyzed (Participants) | 27
hours
  rFVIIIFc Baseline | 0.55 [0.41 to 0.75]
  Advate | 0.46 [0.35 to 0.61]

28. Secondary Outcome: Area Under the Curve (AUC) Per Dose (Two-stage Chromogenic Assay)
Description: as for outcome 7
Time Frame: See Measure Description for complete time frame.
Population: Participants who had evaluable two-stage PK profiles for both Advate and baseline rFVIIIFc.
Measure: Geometric Mean (95% Confidence Interval); unit: IU*h/dL per IU/kg
Arm/Group | Individualized (Tailored) Prophylaxis: Sequential PK Subgroup
Number analyzed (Participants) | 27
IU*h/dL per IU/kg
  rFVIIIFc Baseline | 47.45 [41.55 to 54.18]
  Advate | 28.05 [24.85 to 31.65]

29. Secondary Outcome: Elimination Half Life (t1/2; Two-stage Chromogenic Assay)
Description: as for outcome 8
Time Frame: See Measure Description for complete time frame.
Population: Participants who had evaluable two-stage PK profiles for both Advate and baseline rFVIIIFc.
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Individualized (Tailored) Prophylaxis: Sequential PK Subgroup
Number analyzed (Participants) | 27
hours
  rFVIIIFc Baseline | 20.89 [18.23 to 23.93]
  Advate | 13.67 [12.31 to 15.18]

30. Secondary Outcome: Clearance (CL; Two-stage Chromogenic Assay)
Description: as for outcome 9
Time Frame: See Measure Description for complete time frame.
Population: Participants who had evaluable two-stage PK profiles for both Advate and baseline rFVIIIFc.
Measure: Geometric Mean (95% Confidence Interval); unit: mL/h/kg
Arm/Group | Individualized (Tailored) Prophylaxis: Sequential PK Subgroup
Number analyzed (Participants) | 27
mL/h/kg
  rFVIIIFc Baseline | 2.108 [1.846 to 2.407]
  Advate | 3.566 [3.159 to 4.024]

31. Secondary Outcome: Mean Residence Time (MRT; Two-stage Chromogenic Assay)
Description: as for outcome 10
Time Frame: See Measure Description for complete time frame.
Population: Participants who had evaluable two-stage PK profiles for both Advate and baseline rFVIIIFc.
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Individualized (Tailored) Prophylaxis: Sequential PK Subgroup
Number analyzed (Participants) | 27
hours
  rFVIIIFc Baseline | 24.96 [22.41 to 27.80]
  Advate | 15.94 [14.70 to 17.27]

32. Secondary Outcome: Incremental Recovery (Two-stage Chromogenic Assay)
Description: as for outcome 11
Time Frame: See Measure Description for complete time frame.
Population: Participants who had evaluable two-stage PK profiles for both Advate and baseline rFVIIIFc.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL per IU/kg
Arm/Group | Individualized (Tailored) Prophylaxis: Sequential PK Subgroup
Number analyzed (Participants) | 27
IU/dL per IU/kg
  rFVIIIFc Baseline | 2.4912 [2.2762 to 2.7265]
  Advate | 2.5589 [2.3247 to 2.8168]

33. Secondary Outcome: Hemophilia-Specific Quality of Life Index for Adults (Haem-A-QoL) Questionnaire: Change From Baseline to Week 14
Description: The Haem-A-QoL consists of items pertaining to 10 domains specific to living with hemophilia and was administered to adult participants (17 years and older). The 10 domains are: physical health, feeling, view of yourself, sports/leisure, school/work, dealing with hemophilia, and treatment (time frame for all 7 domains, during the last month) and future, family planning, and outlook for the future (time frame for all 3 domains, recently). Lower scores represent better QoL; therefore, a negative change from baseline represents improvement during the course of the study. Scores on a scale range between 0 and 100. Participants in Arm 1 were stratified by their prestudy regimen (either prophylaxis or on-demand).
Time Frame: Baseline, Week 14
Population: Full Analysis Set: participants over 17 years of age who received at least 1 dose of rFVIIIFc and had an assessment. n=participants who had specified assessment at given timepoint.
Measure: Median (Full Range); unit: units on a scale
Groups:
- Arm 1: Individualized Prophylaxis, Prestudy Prophylaxis; Arm 1: Individualized Prophylaxis, Prestudy On-demand: On rFVIIIFc Day 0, all participants underwent pharmacokinetic (PK) analysis with 50 IU/kg rFVIIIFc to estimate their PK parameters and guide the appropriate dose or interval of dosing. A subset of participants (Sequential PK subgroup) also had PK analyses performed with a single dose of 50 IU/kg Advate (Advate Day 0) within 8 weeks prior to rFVIIIFc Day 0. A >= 96 hour washout was performed before the PK dose of Advate or rFVIIIFc was administered. Repeat PK profiling with a single dose of 50 IU/kg rFVIIIFc was conducted at Week 14 or after 12 to 24 weeks of prophylaxis with rFVIIIFc.
  After PK assessments, all participants started twice weekly treatment with 25 IU/kg of rFVIIIFc via intravenous (IV) injection on Day 1 and 50 IU/kg on Day 4, followed by individualized dose and interval modification within the range of 25 to 65 IU/kg every 3 to 5 days, as determined by rFVIIIFc PK analysis, to maintain a trough level of 1% to 3% (or higher, as clinically indicated) FVIII activity.
Arm/Group | Arm 1: Individualized Prophylaxis, Prestudy Prophylaxis | Arm 1: Individualized Prophylaxis, Prestudy On-demand | Arm 2: Weekly Prophylaxis | Arm 3: Episodic (On-Demand) Dosing
Number analyzed (Participants) | 69 | 22 | 15 | 17
units on a scale
  Total Score (n=57, 17, 14, 14) | -2.18 [-25.0 to 20.9] | -1.48 [-28.6 to 5.1] | -4.73 [-30.5 to 3.2] | -2.09 [-25.1 to 5.4]
  Physical Health (n=68, 22, 15, 17) | -5.00 [-70.0 to 75.0] | -12.50 [-42.5 to 45.0] | -10.0 [-40.0 to 10.0] | 0.00 [-55.0 to 40.0]
  Feeling (n=68, 22, 15, 17) | 0.00 [-43.8 to 43.8] | -6.25 [-37.5 to 12.5] | -6.25 [-50.0 to 6.3] | -6.25 [-37.5 to 6.3]
  View of Yourself (n=68, 22, 15, 17) | 0.00 [-70.0 to 25.0] | 5.00 [-30.0 to 25.0] | 0.00 [-30.0 to 15.0] | -5.00 [-40.0 to 20.0]
  Sports and Leisure (n=48, 12, 12, 8) | 0.00 [-55.0 to 40.0] | -2.50 [-25.0 to 18.8] | -10.0 [-30.0 to 0.0] | -2.50 [-30.0 to 15.0]
  Work and School (n=53, 17,13, 14) | -6.25 [-56.3 to 25.0] | -6.25 [-37.5 to 25.0] | 0.00 [-31.3 to 39.6] | 0.00 [-58.3 to 12.5]
  Dealing with Hemophilia (n=65, 22, 15, 17) | 0.00 [-33.3 to 50.0] | 0.00 [-25.0 to 16.7] | 0.00 [-25.0 to 41.7] | 0.00 [-50.0 to 100.0]
  Treatment (n=68, 21, 15, 16) | -3.13 [-37.1 to 21.9] | -3.13 [-43.8 to 31.3] | -3.13 [-31.3 to 18.8] | 0.00 [-21.9 to 18.8]
  Future (n=66, 21, 15, 17) | 2.50 [-35.0 to 25.0] | 0.00 [-30.0 to 55.0] | -5.00 [-35.0 to 15.0] | -5.00 [-55.0 to 25.0]
  Family Planning (n=38, 10, 8, 7) | 0.00 [-31.3 to 18.8] | 0.00 [-18.8 to 31.3] | 0.00 [-50.0 to 8.3] | -2.08 [-31.3 to 0.0]
  Partnership and Sexuality (n=62, 20, 15, 17) | 0.00 [-25.0 to 41.7] | 0.00 [-25.0 to 58.3] | 0.00 [-41.7 to 0.0] | 0.00 [-100.0 to 25.0]

34. Secondary Outcome: Hemophilia-Specific Quality of Life Index for Adults (Haem-A-QoL) Questionnaire: Change From Baseline to Week 28
Description: as for outcome 33
Time Frame: Baseline, Week 28
Population: as for outcome 33
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Arm 1: Individualized Prophylaxis, Prestudy Prophylaxis | Arm 1: Individualized Prophylaxis, Prestudy On-demand | Arm 2: Weekly Prophylaxis | Arm 3: Episodic (On-Demand) Dosing
Number analyzed (Participants) | 42 | 17 | 3 | 7
units on a scale
  Total Score (n=34, 12, 3, 5) | -1.03 [-26.7 to 11.5] | -4.31 [-35.6 to 13.9] | -5.81 [-9.8 to 5.4] | -0.56 [-11.2 to 3.4]
  Physical Health (n=40, 17, 3, 7) | 0.00 [-31.3 to 60.0] | -25.00 [-65.0 to 25.0] | -5.00 [-45.0 to -5.0] | 0.00 [-15.0 to 20.0]
  Feeling (n=40, 17, 3, 7) | -3.13 [-50.0 to 25.0] | -6.25 [-50.0 to 18.8] | -6.25 [-18.8 to 6.3] | 0.00 [-12.5 to 18.8]
  View of Yourself (n=42, 17, 3, 7) | 0.00 [-40.0 to 35.0] | 0.00 [-40.0 to 20.0] | 0.00 [-5.0 to 5.0] | 0.00 [-5.0 to 15.0]
  Sports and Leisure (n=29, 10, 2, 5) | 0.00 [-68.8 to 45.0] | -5.00 [-50.0 to 5.0] | -10.0 [-25.0 to 5.0] | 5.00 [-8.8 to 5.0]
  Work and School (n=34, 15, 2, 6) | 0.00 [-50.0 to 37.5] | -6.25 [-56.3 to 25.0] | -9.38 [-18.8 to 0.0] | -3.13 [-25.0 to 6.3]
  Dealing with Hemophilia (n=40, 17, 3, 7) | 0.00 [-33.3 to 33.3] | 0.00 [-25.0 to 58.3] | 0.00 [-16.7 to 25.0] | 0.00 [-16.7 to 8.3]
  Treatment (n=42, 14, 3, 7) | 0.00 [-28.1 to 18.8] | -4.69 [-43.8 to 12.5] | 6.25 [-12.5 to 28.1] | 0.00 [-18.8 to 6.3]
  Future (n=40, 17, 3, 6) | 0.00 [-45.0 to 35.0] | -5.00 [-45.0 to 60.0] | -5.00 [-20.0 to -5.0] | 7.50 [-15.0 to 10.0]
  Family Planning (n=19, 10, 2, 2) | 0.00 [-25.0 to 16.7] | 0.00 [-18.8 to 33.3] | 0.00 [0.0 to 0.0] | 9.38 [0.0 to 18.8]
  Partnership and Sexuality (n=37, 14, 3, 7) | 0.00 [-25.0 to 66.7] | 0.00 [-25.0 to 91.7] | 0.00 [-8.3 to 0.0] | 0.00 [-25.0 to 8.3]

35. Secondary Outcome: Hemophilia-Specific Quality of Life Index for Children (Haemo-QoL) Questionnaire: Change From Baseline to Week 14 and Week 28 in Haemo-QoL III Total Score
Description: The Haemo-QoL III, a quality of life assessment instrument for adolescents with hemophilia, was administered to participants from 13 to 16 years old. This instrument assesses domains specific to living with hemophilia and consists of 12 domains: physical health, feeling, view of yourself, family, friends, others, sports and school, treatment, perceived support, dealing with hemophilia, future, and relationships. Total HAEMO-QoL score is the sum of all raw scores for all subscales for participants for whom at least the minimum number of required questions have been answered. Total scores are presented as the Transformed Scale Score (TSS) from 0-100%, with lower scores indicating a better quality of life. A negative change indicates improvement.
Time Frame: Baseline, Week 14, Week 28
Population: Full Analysis Set: participants 13 to 16 years of age who received at least 1 dose of rFVIIIFc and had an assessment. n=participants who had specified assessment at given timepoint.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Arm 1: Individualized (Tailored) Prophylaxis | Arm 2: Weekly Prophylaxis | Arm 3: Episodic (On-Demand) Dosing
Number analyzed (Participants) | 8 | 0 | 2
units on a scale
  Baseline (n=8, 0, 2) | 11.20 [6.5 to 38.3] |  | 26.30 [16.2 to 36.4]
  Change from Baseline at Week 14 (n=8, 0, 1) | -3.25 [-21.9 to 2.3] |  | -5.01 [-5.01 to -5.01]
  Change from Baseline at Week 28 (n=4, 0, 0) | -3.73 [-6.2 to -1.3] |  | NA [NA to NA] — n=0 for this timepoint

36. Secondary Outcome: Investigators'/Surgeons' Assessment of Participants' Response to rFVIIIFc for Major Surgery
Description: Based on the first assessment of hemostasis by the surgeon/investigator 24 hours or later post-surgery. Scaled responses: Excellent = 1, Good = 2, Fair = 3, Poor/none = 4.
Time Frame: up to 52 weeks
Population: Participants in the Full Analysis Set (FAS) who received at least 1 dose of rFVIIIFc and underwent major surgery.
Measure: Number; unit: responses
Units Other Than Participants: Major Surgeries
Groups:
- Perioperative Management (Surgery) Subgroup: Participants from any arm who underwent major surgery. The surgical period and dosing were dependent on the type of surgery the participant underwent.
Arm/Group | Perioperative Management (Surgery) Subgroup
Number analyzed (Participants) | 9
Number analyzed (Major Surgeries) | 9
responses
  Excellent or Good | 9
  Excellent | 8
  Good | 1
  Fair | 0
  Poor/None | 0

37. Secondary Outcome: Number of Injections Required to Maintain Hemostasis During Major Surgery
Description: The number of injections to maintain hemostasis during surgery includes all injections for surgery purposes, including from the loading dose to the end date/time of surgery.
Time Frame: up to 52 weeks
Population: Participants in the Full Analysis Set (FAS) who received at least 1 dose of rFVIIIFc and underwent major surgery.
Measure: Median (Full Range); unit: injections
Units Other Than Participants: Major Surgeries
Arm/Group | Perioperative Management (Surgery) Subgroup
Number analyzed (Participants) | 9
Number analyzed (Major Surgeries) | 9
injections | 1.0 [1 to 1]

38. Secondary Outcome: Dose Per Injection and Total Dose Required to Maintain Hemostasis During Major Surgery
Description: Mean dose per injection is the average dose for all injections (including loading dose) needed to maintain hemostasis during surgery. Total dose is the sum across all injections (including loading dose) needed to maintain hemostasis during surgery.
Time Frame: up to 52 weeks ± 2 weeks
Population: Participants in the Full Analysis Set (FAS) who received at least 1 dose of rFVIIIFc and underwent major surgery.
Measure: Median (Full Range); unit: IU/kg
Units Other Than Participants: Major Surgeries
Arm/Group | Perioperative Management (Surgery) Subgroup
Number analyzed (Participants) | 9
Number analyzed (Major Surgeries) | 9
IU/kg
  Dose per Injection | 51.4 [50 to 77]
  Total Dose | 51.4 [50 to 77]

39. Secondary Outcome: Estimated Total Blood Loss During Major Surgery
Time Frame: up to 52 weeks ± 2 weeks
Population: Participants in the Full Analysis Set (FAS) who received at least 1 dose of rFVIIIFc, underwent major surgery, and had blood loss during surgery information available.
Measure: Median (Full Range); unit: mL
Units Other Than Participants: Major Surgeries
Arm/Group | Perioperative Management (Surgery) Subgroup
Number analyzed (Participants) | 9
Number analyzed (Major Surgeries) | 7
mL | 15.0 [0 to 600]

40. Secondary Outcome: Number of Transfusions Required Per Surgery
Description: Number of blood component transfusions during a single surgery.
Time Frame: up to 52 weeks ± 2 weeks
Population: Participants in the Full Analysis Set (FAS) who received at least 1 dose of rFVIIIFc and underwent major surgery.
Measure: Number; unit: surgeries
Units Other Than Participants: Major Surgeries
Arm/Group | Perioperative Management (Surgery) Subgroup
Number analyzed (Participants) | 9
Number analyzed (Major Surgeries) | 9
surgeries
  0 transfusions | 8
  1 transfusion | 0
  2 transfusions | 1
  3 transfusions | 0
  > 3 transfusions | 0

ADVERSE EVENTS:
Time Frame: up to 52 weeks + 30 days ± 1 week
Description: Based on participants treated with rFVIIIFc in each arm. One participant in Individualized (Tailored) Prophylaxis arm received only Advate and was not included in the treatment-emergent AE table. Does not include SAEs emergent during surgical/rehabilitation period (see Outcome Measure 2 for a summary of treatment-emergent events for this subgroup).
Groups:
- Individualized (Tailored) Prophylaxis, rFVIIIFc: Initial twice weekly dosing with 25 IU/kg of rFVIIIFc via intravenous (IV) injection on Day 1 and 50 IU/kg on Day 4, followed by individualized dose and interval modification within the range of 25 to 65 IU/kg every 3 to 5 days to maintain a trough level of 1% to 3% (or higher, as clinically indicated) rFVIIIFc activity.
  Prior to rFVIIIFc treatment, on rFVIIIFc Day 0, all participants underwent pharmacokinetic (PK) analysis with rFVIIIFc in order to estimate participant's PK parameters and guide the appropriate dose or interval of dosing. Repeat PK profiling with a single dose of 50 IU/kg rFVIIIFc was conducted at Week 14 or after 12 to 24 weeks of prophylaxis with rFVIIIFc.
  A subset of participants (Sequential PK Subgroup) also had PK profiling performed with a single dose of 50 IU/kg Advate (Advate Day 0) within 8 weeks prior to rFVIIIFc Day 0. A >= 96 hour washout from Advate or any other FVIII product was performed before the first PK dose of rFVIIIFc was administered.
- Episodic (On-Demand) Dosing: Initial single dose of 50 IU/kg of rFVIIIFc via IV injection followed by 10 to 50 IU/kg rFVIIIFc, as required to treat a bleeding episode
Arm/Group | Individualized (Tailored) Prophylaxis, rFVIIIFc | Weekly Prophylaxis | Episodic (On-Demand) Dosing
Serious Adverse Events (participants affected / at risk) | 10/117 | 2/24 | 0/23
Other Adverse Events (participants affected / at risk) | 32/117 | 8/24 | 7/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Individualized (Tailored) Prophylaxis, rFVIIIFc (N=117) | Weekly Prophylaxis (N=24) | Episodic (On-Demand) Dosing (N=23)
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypertensive emergency (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Individualized (Tailored) Prophylaxis, rFVIIIFc (N=117) | Weekly Prophylaxis (N=24) | Episodic (On-Demand) Dosing (N=23)
Nasopharyngitis (Infections and infestations) | 16 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 6 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 2 | 1
Headache (Nervous system disorders) | 5 | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.